CLINICAL TRIAL: NCT01795859
Title: A Randomized Double-Blind, Placebo-Controlled Study of SD-809 Extended Release for the Treatment of Chorea Associated With Huntington Disease
Brief Title: First Time Use of SD-809 in Huntington Disease
Acronym: First-HD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SD-809-C-15
Record Dates: First submitted 2013-02-20; First posted 2013-02-21 (Estimated); Results first posted 2017-08-11 (Actual); Last update posted 2017-09-20 (Actual); Status verified 2017-08

CONDITIONS: Chorea
Keywords: Huntington disease; Chorea; Tetrabenazine
MeSH Terms: conditions — Chorea; Huntington Disease | interventions — deutetrabenazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SD-809 ER Tablets (Experimental): SD-809 ER tablets are available in three dose strengths: 6, 9 and 12 mg, all of which are identical in size, shape and color (white). All are administered three times a day, with the 6 mg final dose is placebo.
  Interventions: Drug: SD-809; Drug: Placebo
- SD-809 Tablets (Experimental): SD-809 tablets are available in three dose strengths: 6, 9 and 12 mg, all of which are identical in size, shape and color (white). All are administered three times a day, with the 6 mg final dose is placebo.
  Interventions: Drug: SD-809; Drug: Placebo

INTERVENTIONS:
Drug: SD-809 — SD-809 tablets are available in three dose strengths: 6, 9 and 12 mg, all of which are identical in size, shape and color (white).
  Other Names: deutetrabenazine
Drug: Placebo — Placebo tablets are identical in appearance to SD-809 tablets.

SUMMARY:
The purpose of this study is to determine whether SD-809 tablets are effective in the treatment of chorea associated with Huntington's Disease.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel-group study designed to evaluate the efficacy, safety and tolerability of SD-809 for the treatment of chorea associated with Huntington's Disease. Approximately 90 subjects will be randomized (1:1) into the study, with approximately 45 subjects receiving SD-809 and 45 subjects receiving placebo. The study will be conducted at approximately 30 centers in the U.S. and Canada.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age or the age of majority (whichever is older) at Screening.
* Subject has been diagnosed with manifest HD
* Subject is able to swallow study medication whole.
* Female subjects of childbearing potential agree to use an acceptable method of contraception from screening through study completion.
* The subject has a reliable caregiver who interacts with the patient on a daily basis, oversees study drug administration, assures attendance at study visits and participates in evaluations, as required.
* Subject is able to ambulate without assistance for at least 20 yards (Note: The use of assistive devices (i.e., walker, cane) is permitted during ambulation).

Exclusion Criteria:

* Subject has a serious untreated or under-treated psychiatric illness, such as depression, at Screening or Baseline.
* Subject has active suicidal ideation at Screening or Baseline.
* Subject has history of suicidal behavior at Screening or Baseline:
* Subject has evidence for depression at Screening or Baseline.
* Subject has an unstable or serious medical or psychiatric illness at Screening or Baseline.
* Subject has been recently exposed to tetrabenazine.
* Subject has received any of the following concomitant medications within 30 days of Screening or Baseline:

  * Antipsychotics
  * Metoclopramide
  * Monoamine oxidase inhibitors (MAOI)
  * Levodopa or dopamine agonists
  * Reserpine
  * Amantadine
  * Memantine
* Subject has significantly impaired swallowing function at Screening.
* Subject has significantly impaired speaking at Screening.
* Subject requires treatment with drugs known to prolong the QT interval.
* Subject has a prolonged QT interval on 12-lead ECG at Screening.
* Subject has evidence of hepatic impairment at Screening.
* Subject has evidence of significant renal impairment at Screening.
* Subject has known allergy to any of the components of study medication.
* Subject has participated in an investigational drug or device trial within 30 days (or 5 drug half-lives) of Screening, whichever is longer.
* Subject is pregnant or breast-feeding at Screening or Baseline.
* Subject acknowledges present use of illicit drugs at Screening.
* Subject has a history of alcohol or substance abuse in the previous 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-08-05 (Actual); Primary Completion 2014-12-05 (Actual); Study Completion 2014-12-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (43):
- United States (37):
  - Teva Investigational Site 057, Birmingham, Alabama
  - Teva Investigational Site 038, Phoenix, Arizona
  - Teva Investigational Site 298, Fayetteville, Arkansas
  - Teva Investigational Site 050, Los Angeles, California
  - Teva Investigational Site 052, Englewood, Colorado
  - Teva Investigational Site 333, Washington D.C., District of Columbia
  - Teva Investigational Site 196, Boca Raton, Florida
  - Teva Investigational Site 160, Gainesville, Florida
  - Teva Investigational Site 014, Miami, Florida
  - Teva Investigational Site 032, Atlanta, Georgia
  - Teva Investigational Site 045, Indianapolis, Indiana
  - Teva Investigational Site 024, Iowa City, Iowa
  - Teva Investigational Site 029, Kansas City, Kansas
  - Teva Investigational Site 083, Wichita, Kansas
  - Teva Investigational Site 087, Louisville, Kentucky
  - Teva Investigational Site 028, Baltimore, Maryland
  - Teva Investigational Site 040, Boston, Massachusetts
  - Teva Investigational Site 027, St Louis, Missouri
  - Teva Investigational Site 194, Las Vegas, Nevada
  - Teva Investigational Site 328, Camden, New Jersey
  - Teva Investigational Site 026, New Brunswick, New Jersey
  - Teva Investigational Site 037, Albany, New York
  - Teva Investigational Site 002, New York, New York
  - Teva Investigational Site 342, Patchogue, New York
  - Teva Investigational Site 119, Durham, North Carolina
  - Teva Investigational Site 089, Cincinnati, Ohio
  - Teva Investigational Site 020, Columbus, Ohio
  - Teva Investigational Site 093, Toledo, Ohio
  - Teva Investigational Site 341, Tulsa, Oklahoma
  - Teva Investigational Site 031, Nashville, Tennessee
  - Teva Investigational Site 007, Houston, Texas
  - Teva Investigational Site 199, Houston, Texas
  - Teva Investigational Site 100, Salt Lake City, Utah
  - Teva Investigational Site 137, Burlington, Vermont
  - Teva Investigational Site 220, Kirkland, Washington
  - Teva Investigational Site 096, Seattle, Washington
  - Teva Investigational Site 104, Milwaukee, Wisconsin
- Australia (2):
  - Teva Investigational Site 144, Kew Vic
  - Teva Investigational Site 054, Sydney
- Canada (4):
  - Teva Investigational Site 098, Montreal
  - Teva Investigational Site 300, North York
  - Teva Investigational Site 231, Ottawa
  - Teva Investigational Site 300, Ottawa

REFERENCES:
- [Derived] Frank S, Testa CM, Goldstein J, Kayson E, Leavitt BR, Oakes D, O'Neill C, Whaley J, Gross N, Chaijale N, Barash S, Gordon MF; Huntington Study Group/ARC-HD Investigators and Coordinators. Safety and Efficacy of Deutetrabenazine at High versus Lower Daily Dosages in the ARC-HD Study to Treat Chorea in Huntington Disease. CNS Drugs. 2025 Feb;39(2):185-195. doi: 10.1007/s40263-024-01139-3. Epub 2025 Jan 18. PMID 39825184
- [Derived] Frank S, Anderson KE, Fernandez HH, Hauser RA, Claassen DO, Stamler D, Factor SA, Jimenez-Shahed J, Barkay H, Wilhelm A, Alexander JK, Chaijale N, Barash S, Savola JM, Gordon MF, Chen M. Safety of Deutetrabenazine for the Treatment of Tardive Dyskinesia and Chorea Associated with Huntington Disease. Neurol Ther. 2024 Jun;13(3):655-675. doi: 10.1007/s40120-024-00600-1. Epub 2024 Apr 1. PMID 38557959
- [Derived] Rodrigues FB, Wild EJ. Huntington's Disease Clinical Trials Corner: February 2018. J Huntingtons Dis. 2018;7(1):89-98. doi: 10.3233/JHD-189001. PMID 29480210
- [Derived] Claassen DO, Carroll B, De Boer LM, Wu E, Ayyagari R, Gandhi S, Stamler D. Indirect tolerability comparison of Deutetrabenazine and Tetrabenazine for Huntington disease. J Clin Mov Disord. 2017 Mar 1;4:3. doi: 10.1186/s40734-017-0051-5. eCollection 2017. PMID 28265459
- [Derived] Huntington Study Group; Frank S, Testa CM, Stamler D, Kayson E, Davis C, Edmondson MC, Kinel S, Leavitt B, Oakes D, O'Neill C, Vaughan C, Goldstein J, Herzog M, Snively V, Whaley J, Wong C, Suter G, Jankovic J, Jimenez-Shahed J, Hunter C, Claassen DO, Roman OC, Sung V, Smith J, Janicki S, Clouse R, Saint-Hilaire M, Hohler A, Turpin D, James RC, Rodriguez R, Rizer K, Anderson KE, Heller H, Carlson A, Criswell S, Racette BA, Revilla FJ, Nucifora F Jr, Margolis RL, Ong M, Mendis T, Mendis N, Singer C, Quesada M, Paulsen JS, Brashers-Krug T, Miller A, Kerr J, Dubinsky RM, Gray C, Factor SA, Sperin E, Molho E, Eglow M, Evans S, Kumar R, Reeves C, Samii A, Chouinard S, Beland M, Scott BL, Hickey PT, Esmail S, Fung WL, Gibbons C, Qi L, Colcher A, Hackmyer C, McGarry A, Klos K, Gudesblatt M, Fafard L, Graffitti L, Schneider DP, Dhall R, Wojcieszek JM, LaFaver K, Duker A, Neefus E, Wilson-Perez H, Shprecher D, Wall P, Blindauer KA, Wheeler L, Boyd JT, Houston E, Farbman ES, Agarwal P, Eberly SW, Watts A, Tariot PN, Feigin A, Evans S, Beck C, Orme C, Edicola J, Christopher E. Effect of Deutetrabenazine on Chorea Among Patients With Huntington Disease: A Randomized Clinical Trial. JAMA. 2016 Jul 5;316(1):40-50. doi: 10.1001/jama.2016.8655. PMID 27380342

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 90 subjects were randomized 1:1 to receive either SD-809 or placebo. All subjects were assessed for capacity to provide informed consent and written informed consent was obtained appropriately
Groups:
- SD-809 Placebo: Placebo: Placebo tablets are identical in appearance to SD-809 tablets.
Period: Overall Study
Arm/Group | SD-809 Tablets | SD-809 Placebo
Started | 45 | 45
Completed | 44 | 43
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SD-809 Tablets | SD-809 Placebo | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Customized [Mean (Standard Deviation); unit: participants]
  SD-809 | 55.4 (10.32) | 52.1 (13.36) | 53.7 (11.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 17 | 40
  Male | 22 | 28 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 5 | 5
  White | 45 | 38 | 83
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Average of Screening and Day 0) in the Average TMC Scores From Weeks 9 & 12
Description: Total TMC score is a sum of chorea scores which range 0-28, with a decrease indicating improvement in chorea
Time Frame: Screening, Day 0, Weeks 9, 12
Population: The Modified ITT (mITT) Population was defined as all subjects in the ITT Population who received study drug and had at least one postbaseline assessment. For subjects who missed both Week 9 or Week 12 scores, the last available assessment was used
Measure: Least Squares Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SD-809 Tablets | SD-809 Placebo
Number analyzed (Participants) | 45 | 45
Units on a scale | -4.42 (2.953) | -1.93 (2.666)
Statistical Analysis 1: Comparison: SD-809 Tablets vs SD-809 Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; LSMean Difference = -2.49, 95% CI 2-sided [-3.69 to -1.29]

2. Secondary Outcome: Number of Participants With Treatment Success at the End of Therapy as Measured by the Patient Global Impression of Change (PGIC)
Description: A treatment success is defined as Much or Very Much Improved at the Week 12 visit. The PGIC is a 7-point Likert Scale, ranging from very much worse to very much improved
Time Frame: 12 weeks
Population: The Modified ITT (mITT) Population was defined as all subjects in the ITT Population who received study drug and had at least one post baseline assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | SD-809 Tablets | SD-809 Placebo
Number analyzed (Participants) | 45 | 45
Participants | 23 | 9
Statistical Analysis 1: Comparison: SD-809 Tablets vs SD-809 Placebo; Test type: Superiority or Other; p = 0.0020, Difference of proportions; Mean Difference (Final Values) = 31.1, 95% CI 2-sided [12.4 to 49.8]

3. Secondary Outcome: Number of Participants With Treatment Success at the End of Therapy Based on Clinical Global Impression of Change (CGIC)
Description: A treatment success is defined as Much or Very Much Improved at the Week 12 visit. The PGIC is a 7-point Likert Scale, ranging from very much worse to very much improved. The clinician was asked to comment about the subject.
Time Frame: 12 weeks
Population: The Modified ITT (mITT) Population was defined as all subjects in the ITT Population who received study drug and had at least one post-baseline assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | SD-809 Tablets | SD-809 Placebo
Number analyzed (Participants) | 45 | 45
Participants | 19 | 6
Statistical Analysis 1: Comparison: SD-809 Tablets vs SD-809 Placebo; Test type: Superiority or Other; p = 0.0022, Difference of proportions; Mean Difference (Final Values) = 28.9, 95% CI 2-sided [11.4 to 46.4]

4. Secondary Outcome: Change in the Short Form 36 Health Survey (SF-36) Physical Functioning Score (Based on Items 3a to 3j) From Baseline to Week 12
Description: Change in the Short Form 36 Health Survey (SF-36) physical functioning score (based on items 3a to 3j) from Baseline to Week 12. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Time Frame: Baseline, 12 weeks
Population: The modified intent to treat (mITT) population will include all subjects in the ITT population who were randomized to treatment and received study drug. For subjects with missing value at Week 12, the last available assessment was used
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SD-809 Tablets | SD-809 Placebo
Number analyzed (Participants) | 45 | 43
units on a scale | 0.74 (9.773) | -3.61 (9.669)
Statistical Analysis 1: Comparison: SD-809 Tablets vs SD-809 Placebo; Test type: Superiority or Other; p = 0.0308, Mixed Models Analysis; LSMean Difference = 4.34, 95% CI 2-sided [0.41 to 8.27]

5. Secondary Outcome: Change in Berg Balance Test (BBT)
Description: The Berg Balance Test (BBT) is a 14-item assessment of sitting, standing, transferring, and turning. Each task ranging from standing up from a sitting position, to standing on one foot each task is given a score of zero (unable) to four (independent), and the final measure is the sum of all of the scores.The scale range, which is 0-56, with higher scores indicating better balance/lower fall risk.
Time Frame: Baseline, 12 weeks
Population: The Modified ITT (mITT) Population was defined as all subjects in the ITT Population who received study drug and had at least one postbaseline assessment. For subjects with missing value at Week 12, the last available assessment was used
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | SD-809 Tablets | SD-809 Placebo
Number analyzed (Participants) | 45 | 45
units on a scale | 2.2 (3.47) | 1.3 (4.04)
Statistical Analysis 1: Comparison: SD-809 Tablets vs SD-809 Placebo; Test type: Superiority or Other; p = 0.1415, Mixed Models Analysis; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [-0.3 to 2.3]

ADVERSE EVENTS:
Groups:
- Placebo: Placebo
- SD-809: SD-809
Arm/Group | Placebo | SD-809
Serious Adverse Events (participants affected / at risk) | 1/45 | 1/45
Other Adverse Events (participants affected / at risk) | 21/45 | 18/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=45) | SD-809 (N=45)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Agitated depression (Psychiatric disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=45) | SD-809 (N=45)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 4 (4)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Fatigue (General disorders) | 2 (2) | 3 (4)
Irritability (General disorders) | 6 (6) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 4 (6) | 2 (4)
Dizziness (Nervous system disorders) | 4 (4) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 5 (6)
Depression (Psychiatric disorders) | 3 (3) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 3 (3)
Sleep disorder (Psychiatric disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less